CLINICAL TRIAL: NCT03056170
Title: Neurophysiological Impact of a Fronto-temporal Transcranial Direct Current Stimulation (tDCS) in Healthy Subjects: a Multimodal Imaging Approach
Brief Title: Neurophysiological Impact of a Fronto-temporal tDCS Stimulation in Healthy Subjects: a Multimodal Imaging Approach
Acronym: COMBI-STIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 69HCL16_0682
Record Dates: First submitted 2017-02-08; First posted 2017-02-17 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS (Active Comparator): The anode is placed over the left dorsolateral prefrontal cortex (DLPFC) and the cathode is placed over the left temporo-parietal cortex (TPJ) In active stimulation with a Transcranial Direct Current Stimulation, the device will deliver a charge of 1 mA for 30 minutes.
  Interventions: Device: real tDCS
- Sham tDCS (Sham Comparator): In sham stimulation, with a Transcranial Direct Current Stimulation, no current will be delivered from one electrode to the other except one 30 s ramp up and down at the beginning and one at the end of the sham stimulation duration (30 min) Same electrode montage than in the active group.
  Interventions: Device: real tDCS

INTERVENTIONS:
Device: real tDCS — In active stimulation, the "Transcranial Direct Current Stimulation" device will produce a direct current of 1 mA from one electrode to the other for 30 min with a ramp up at the beginning and a ramp down at the end of the stimulation of 30 s. The sham or active mode is chosen by a numeric code.

SUMMARY:
tDCS is a technique emerging as a prospective therapy for neurologic, psychiatric and addictive disorders. Specifically, fronto-temporal tDCS, with anodal stimulation over the left dorsolateral prefrontal cortex (DLPFC) and cathodal stimulation over the left temporo-parietal junction (TPJ), has been reported to reduce treatment-resistant auditory hallucinations (AH), negative symptoms and insight of the illness in schizophrenia. However, despite an increasing use in clinical settings, tDCS suffers from limitations, especially regarding the strength and the duration of therapeutic effects.

Some imaging reports suggest that tDCS effects are not restricted to the brain areas located under the electrodes, but spread through distributed cortical networks functionally connected with the targets and reach subcortical areas. Overall, these studies suggest that tDCS modulates functional connectivity within and across resting-state networks and brain activity. However, these effects are currently described at different levels depending on the imaging technique used. Moreover, the majority of studies have focused on motor cortex stimulation, while the specific effects of fronto-temporal tDCS are scarce. Finally, effects of the stimulation applied online are rarely inspected.

According to the therapeutic effects of fronto-temporal tDCS on schizophrenia and the dopaminergic pathophysiological hypothesis of schizophrenia, the effect of fronto-temporal tDCS on dopaminergic transmission is of major interest. As the cortex is densely connected with basal ganglia areas, tDCS effects are probably capable to reach subcortical dopaminergic areas. Indeed, recent fMRI studies highlighted subcortical effects of tDCS applied at the cortical level including modulations of cortico-striatal and thalamo-cortical functional connectivity. In addition, some studies suggest that cortical stimulation by other approaches, such as transcranial magnetic stimulation (rTMS) modulates dopaminergic transmission. However, tDCS effects on dopaminergic transmission have been investigated only indirectly.

Finally, information about biological effects of tDCS is scattered and creating a coherent ensemble is a mandatory and critical step to understand the mechanisms of action of tDCS.

According to the hypothesis that fronto-temporal tDCS modulates brain activity, connectivity and dopaminergic transmission, the aim of this project is to reveal the combined neurobiological impact of an online single session of fronto-temporal tDCS in a unique experiment by developing a simultaneous multimodal imaging approach (PET-MRI). The online implementation of the stimulation will allow deciphering changes induced during and after stimulation. As a first step before investigating patients with schizophrenia, healthy subjects will be involved in the present study.

The distributed changes will be explored at rest through:

* Spontaneous functional connectivity assessed by functional magnetic resonance imagery (fMRI).
* Brain activity assessed by cerebral blood flow quantitatively and directly measured by arterial spin labelling (ASL).
* Connectivity assessed by diffusion tensor imaging (DTI).
* Specific and localized dopaminergic transmission evaluated by positron emission tomography (PET) using dopaminergic D2 subtype receptor availability via [11C]raclopride binding.

The pioneering aspects of the project are to use an innovative simultaneous multimodal imaging system, adopt the tDCS montage used in our validated therapeutic context and apply tDCS online. We expect that our unique approach will provide an imaging biomarker essential to improve our understanding of:

1. the "normal brain" and further deficient mechanisms underlying schizophrenia as well as neurological disorders.
2. neurobiological effects of tDCS in order to:

   * Bring key element of the proof of concept of tDCS
   * Optimize tDCS in a therapeutic context
   * Suggest a marker of the therapeutic response

ELIGIBILITY:
Inclusion Criteria:

* non smoker
* right handed
* non psychotropic consumption
* no medical treatment except oral contraception
* no psychiatric or somatic (neurological, endocrine, cardiac, renal) disorders
* affiliated to the French social security

Exclusion Criteria:

* No Consent formed signed
* For female participants : pregnancy
* contraindications to stimulation by tDCS or to an MRI exam
* being in an exclusion period or over the annual compensation threshold
* participation in another study using ionizing radiation in less than a year

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Change in dopamine transmission induced by 1 session of 30min tDCS | Continuous measure during 110min of PET scan
  Measure of the Binding Ratio of the radiomarker defined as the ratio of : region of interest / cerebellum activities

SECONDARY OUTCOMES:
Change in spontaneous functional connectivity (using rs fMRI) during and after 1 session of 30min tDCS | - Before stimulation : t+15 to t+28min - During stimulation : t+45 to t+58min - After stimulation : t+76 to t+89min
  The impact of tDCS will be analysed using functional connectivity maps seeded from stimulated regions and from areas belonging to specific networks. Data will be preprocessed and analyzed using specific toolbox.
Change in cerebral blood flow (using ASL) during and after 1 session of 30min tDCS | - Before stimulation : t+30 to t+36min - During stimulation : t+60 to t+66min - After stimulation : t+91 to t+97min
  The impact of tDCS will be analysed using quantitative CBF maps seeded from stimulated regions and from areas belonging to specific networks. Data will be preprocessed and analyzed using specific toolbox.
Change in structural connectivity (using DTI) after 1 session of 30min tDCS | - Before stimulation : t+0 to t+10min - After stimulation : t+100 to t+110min
  The impact of tDCS will be analysed using a tractography-based analysis. Data will be preprocessed and analyzed using specific toolbox.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Haesebaert, MD, Principal Investigator — LE VINATIER
Locations (1):
- Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fonteneau C, Merida I, Redoute J, Haesebaert F, Lancelot S, Costes N, Mondino M, Brunelin J. Modulation of dopaminergic transmission and brain activity by frontotemporal tDCS: A multimodal PET-MR imaging study. Brain Stimul. 2025 Jul-Aug;18(4):1065-1073. doi: 10.1016/j.brs.2025.05.006. Epub 2025 May 6. PMID 40340023